CLINICAL TRIAL: NCT02532400
Title: Comparison of Neoadjuvant Aromatase Inhibitors With Ovarian Suppression Versus Chemotherapy in Premenopausal Patients With Hormone Receptor-positive Breast Cancer (COMPETE): a Randomized Phase 3 Trial
Brief Title: Neoadjuvant Aromatase Inhibitor(AI) With Ovarian Suppression Versus Chemotherapy in Premenopausal Breast Cancer Patients
Acronym: COMPETE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Hard to enroll expected number of eligible patients.
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Li Zhu, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJBC1505
Record Dates: First submitted 2015-08-17; First posted 2015-08-25 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: Breast Neoplasms; Neoadjuvant Endocrine Therapy; Ovarian Function Suppression; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoadjuvant endocrine therapy (Experimental): Six months of exemestane or anastrozole plus goserelin.
  Interventions: Drug: Neoadjuvant endocrine therapy
- Neoadjuvant chemotherapy (Active Comparator): Six cycles of docetaxel plus epirubicin and cyclophosphamide(TEC).
  Interventions: Drug: Neoadjuvant chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant endocrine therapy — Goserelin: 3.6mg, d1, hypodermic injection , q28d*7 plus exemestane: 25mg, po, qd*24w, or anastrozole: 1mg, po, qd*24w
  Other Names: Goserelin and AI
  Arms: Neoadjuvant endocrine therapy
Drug: Neoadjuvant chemotherapy — Docetaxel: 75mg/m2, d1, q3w*6, Epirubicin 75mg/m2, d1, q3w*6 and Cyclophosphamide: 500mg/m2, d1, q3w*6
  Other Names: TEC
  Arms: Neoadjuvant chemotherapy

SUMMARY:
To compare the efficacy and safety of neoadjuvant aromatase inhibitor plus ovarian suppression with chemotherapy in premenopausal patients with hormone receptor-positive breast cancer.

DETAILED DESCRIPTION:
Neoadjuvant therapy is nowadays the standard treatment for both early stage and locally advanced breast cancer, and exhibited similar benefit compared with adjuvant therapy in terms of disease free and overall survival. Patients achieved pathological complete response(pCR) after neoadjuvant chemotherapy have superior outcome compared with those with residual tumors in breast and/or axilla. pCR is now the most wildly accepted surrogate marker for long-term survival of patients, especially in those with triple negative or human epidermal growth factor receptor-2(HER2)-positive breast cancer. However, in luminal HER2-negative breast cancer, neoadjuvant chemotherapy is not as effective as in other subtypes of breast cancer, pCR is less noted and seems barely correlated to long-term survival benefit.

In postmenopausal patients with hormone receptor-positive breast cancer, neoadjuvant endocrine therapy of aromatase inhibitor achieved similar clinical response rate compared with neoadjuvant chemotherapy, and in premenopausal hormone receptor-positive, HER2-negative breast cancer patients, neoadjuvant aromatase inhibitor plus ovarian function suppression(OFS) has showed more pronounced efficacy than tamoxifen plus OFS.

In adjuvant setting, aromatase inhibitor combined with OFS in premenopausal patients with hormone receptor-positive breast cancer has demonstrated superior benefit in terms of disease free survival, and has been established as one of the routine options of adjuvant endocrine therapy. Notwithstanding the remarkable performance of combination of aromatase inhibitor and OFS in adjuvant therapy, the role of this treatment strategy in neoadjuvant setting has yet not been proved when compared with neoadjuvant chemotherapy.

The aim of this study is to prospectively compare the efficacy and safety of neoadjuvant aromatase inhibitor plus OFS with chemotherapy in premenopausal patients with hormone receptor-positive HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Women aged ≥ 18 years
3. Histologically confirmed invasive breast cancer
4. American Joint Committee on Cancer (AJCC) stage: ⅡA-ⅢC, no evidence of metastasis
5. At least one measurable disease in breast and/or axilla
6. ER and/or progesterone receptor(PgR) positive(≥10% of the cells by IHC)
7. HER2 negative(by IHC and/or FISH)
8. Premenopause status (estradiol in premenopausal range or with normal menstrual cycle in the past 6 months with no use of hormonal drugs)
9. Eastern Cooperative Oncology Group（ECOG）score 0-1, an estimated life expectancy of at least 12 months
10. Adequate bone marrow function: Leukocyte ≥ 3.0*109/L; Neutrophil ≥ 1.5*109/L; Hb ≥ 100g/L; Platelet(PLT） ≥ 80*109/L
11. Adequate liver, renal function and coagulation function: Alanine transaminase（ALT） and/or Aspartate transaminase（AST）≤ 1.5 upper normal limit（UNL）, total bilirubin ≤upper normal limit, creatinine ≤ 110umol/L, Creatinine clearance > 60ml/min, blood urea nitrogen（BUN） ≤ 7.1mmol/L, activated partial thromboplastin time（APTT） ≤ 1.5 upper normal limit（UNL）
12. Women with child-bearing potential must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to use an acceptable method of birth control to avoid pregnancy for the duration of the study
13. Serological records of hepatitis B virus（HBV）and hepatitis C virus（HCV） testing.

Exclusion Criteria:

1. Stage IV breast cancer
2. Prior systemic or loco-regional treatment of breast cancer
3. Any anti-neoplastic treatment within 28 days before the beginning of study
4. Known severe hypersensitivity to any drugs in this study
5. History of malignancy within 5 years except carcinoma in situ of cervix or skin basal cell carcinoma that had received adequate treatment
6. Peripheral neuropathy ≥ 2°, according to National Cancer Institute(NCI) Common Terminology Criteria for Adverse Events(CTCAE)(Version 4.0)
7. Any cardiac or pulmonary dysfunction defined as following:

(1) ≥ 3° symptomatic congestive heart failure (CHF) according to NCI CTCAE(Version 4.0) or ≥ 2° CHF according to New York Heart Association（NYHA）

(2) Angina that needs anti-anginal drugs, advanced conduction abnormality or significant vascular disease

(3) Uncontrolled high-risk arrhythmia: atrial tachycardia that silent heart rate >100/min, significant ventricular arrythmia or advanced atrioventricular block(2° type II atrioventricular or 3° atrioventricular block)

(4) Poorly controlled hypertension (systolic BP > 180 mmHg or diastolic BP > 100 mmHg)

(5) Transmural myocardial infarction in EKG

(6) Long-term oxygen therapy

8. Uncontrolled severe systemic disease(clinically significant cardiovascular disease，pulmonary disease or metabolic disease, wound healing disorder, ulcer, severe infection)

9. Pregnant or breast feeding

10. Major operation, obvious trauma within 28 days before randomization or planned major operation during the study

11. Known active hepatic disease due to hepatitis B virus, hepatitis C virus, auto-immune liver disease or sclerosing cholangitis

12. Known HIV infection

13. Any reasons investigators consider that not suitable for the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-03; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate(ORR) | up to 7 months
  Overall response rate(ORR) is defined as complete response rate plus partial response rate.

SECONDARY OUTCOMES:
Pathological complete response(pCR) | up to 7 months
Breast conserving surgery(BCS) rate | up to 7 months
Incidence of neutropenia fever | participants will be followed during the six months of neoadjuvant therapy
Incidence of hot flushes/flashes | participants will be followed during the six months of neoadjuvant therapy
Incidence of osteoporosis | participants will be followed during the six months of neoadjuvant therapy
Incidence of grade 3-4 adverse events | participants will be followed during the six months of neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhu, Prof, Principal Investigator — Comprehensive Breast Health Center, Ruijin Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Coates AS, Winer EP, Goldhirsch A, Gelber RD, Gnant M, Piccart-Gebhart M, Thurlimann B, Senn HJ; Panel Members. Tailoring therapies--improving the management of early breast cancer: St Gallen International Expert Consensus on the Primary Therapy of Early Breast Cancer 2015. Ann Oncol. 2015 Aug;26(8):1533-46. doi: 10.1093/annonc/mdv221. Epub 2015 May 4. PMID 25939896
- [Background] Mauri D, Pavlidis N, Ioannidis JP. Neoadjuvant versus adjuvant systemic treatment in breast cancer: a meta-analysis. J Natl Cancer Inst. 2005 Feb 2;97(3):188-94. doi: 10.1093/jnci/dji021. PMID 15687361
- [Background] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812
- [Background] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Background] Semiglazov VF, Semiglazov VV, Dashyan GA, Ziltsova EK, Ivanov VG, Bozhok AA, Melnikova OA, Paltuev RM, Kletzel A, Berstein LM. Phase 2 randomized trial of primary endocrine therapy versus chemotherapy in postmenopausal patients with estrogen receptor-positive breast cancer. Cancer. 2007 Jul 15;110(2):244-54. doi: 10.1002/cncr.22789. PMID 17538978
- [Background] Ellis MJ, Suman VJ, Hoog J, Lin L, Snider J, Prat A, Parker JS, Luo J, DeSchryver K, Allred DC, Esserman LJ, Unzeitig GW, Margenthaler J, Babiera GV, Marcom PK, Guenther JM, Watson MA, Leitch M, Hunt K, Olson JA. Randomized phase II neoadjuvant comparison between letrozole, anastrozole, and exemestane for postmenopausal women with estrogen receptor-rich stage 2 to 3 breast cancer: clinical and biomarker outcomes and predictive value of the baseline PAM50-based intrinsic subtype--ACOSOG Z1031. J Clin Oncol. 2011 Jun 10;29(17):2342-9. doi: 10.1200/JCO.2010.31.6950. Epub 2011 May 9. PMID 21555689
- [Background] Masuda N, Sagara Y, Kinoshita T, Iwata H, Nakamura S, Yanagita Y, Nishimura R, Iwase H, Kamigaki S, Takei H, Noguchi S. Neoadjuvant anastrozole versus tamoxifen in patients receiving goserelin for premenopausal breast cancer (STAGE): a double-blind, randomised phase 3 trial. Lancet Oncol. 2012 Apr;13(4):345-52. doi: 10.1016/S1470-2045(11)70373-4. Epub 2012 Jan 20. PMID 22265697
- [Background] Pagani O, Regan MM, Walley BA, Fleming GF, Colleoni M, Lang I, Gomez HL, Tondini C, Burstein HJ, Perez EA, Ciruelos E, Stearns V, Bonnefoi HR, Martino S, Geyer CE Jr, Pinotti G, Puglisi F, Crivellari D, Ruhstaller T, Winer EP, Rabaglio-Poretti M, Maibach R, Ruepp B, Giobbie-Hurder A, Price KN, Bernhard J, Luo W, Ribi K, Viale G, Coates AS, Gelber RD, Goldhirsch A, Francis PA; TEXT and SOFT Investigators; International Breast Cancer Study Group. Adjuvant exemestane with ovarian suppression in premenopausal breast cancer. N Engl J Med. 2014 Jul 10;371(2):107-18. doi: 10.1056/NEJMoa1404037. Epub 2014 Jun 1. PMID 24881463
- [Background] Francis PA, Regan MM, Fleming GF, Lang I, Ciruelos E, Bellet M, Bonnefoi HR, Climent MA, Da Prada GA, Burstein HJ, Martino S, Davidson NE, Geyer CE Jr, Walley BA, Coleman R, Kerbrat P, Buchholz S, Ingle JN, Winer EP, Rabaglio-Poretti M, Maibach R, Ruepp B, Giobbie-Hurder A, Price KN, Colleoni M, Viale G, Coates AS, Goldhirsch A, Gelber RD; SOFT Investigators; International Breast Cancer Study Group. Adjuvant ovarian suppression in premenopausal breast cancer. N Engl J Med. 2015 Jan 29;372(5):436-46. doi: 10.1056/NEJMoa1412379. Epub 2014 Dec 11. PMID 25495490